CLINICAL TRIAL: NCT03731026
Title: Evaluation of the LightPath® Imaging System and the PET Tracer 68Ga-RM2 in Wide Local Excision (WLE) for Breast Cancer
Brief Title: The LightPath® and 68Ga-RM2 in Breast Cancer Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lightpoint Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: LPM-008
Record Dates: First submitted 2018-07-25; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — BAY 86-7548

STUDY DESIGN:
Intervention Model Description: 3-Group Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Other): Patient will receive an IV injection of up to 200MBq 68Ga-RM2. Each patient will have torso PET/CT imaging at 2 timepoints. Alternate patients will have imaging at 1 and 2h post-injection then the next patientat 1 and 3h post-injection, with axillary gamma probe measurements (using a collimator) of 68Ga-RM2 at the same time points.
  Interventions: Drug: 68Ga-RM2
- Group 2 (Experimental): WLE will be performed as per standard of care but will also include Intraoperative LightPath® Imaging with 68Ga-RM2. Group 2 scans will acquire LightPath® images of both intact and incised cancer specimens with varying parameters to optimise imaging.
  Interventions: Combination Product: LightPath® Imaging System and 68Ga-RM2
- Group 3 (Experimental): WLE will be performed as per standard of care but will also include Intraoperative LightPath® Imaging with 68Ga-RM2. Group 3 scans will acquire LightPath® images of intact and incised cancer specimens using a final and consistent imaging procedure.
  Interventions: Combination Product: LightPath® Imaging System and 68Ga-RM2

INTERVENTIONS:
Combination Product: LightPath® Imaging System and 68Ga-RM2 — Imaging System:The LightPath® Imaging System is an in vitro diagnostic device which has CE mark in Europe, in line with In Vitro Diagnostic Medical Devices 98/79/EC (post-marketing study).
  Radiopharmaceutical: 68Ga-RM2 is an investigational Positron Emission Tomography (PET)/ Computed Tomography (CT) radiopharmaceutical.
  Arms: Group 2; Group 3
Drug: 68Ga-RM2 — Radiopharmaceutical: 68Ga-RM2 is an investigational Positron Emission Tomography (PET)/ Computed Tomography (CT) radiopharmaceutical.
  Arms: Group 1

SUMMARY:
This study is a prospective, open-label study to examine the performance of the LightPath® Imaging System using the PET tracer 68Ga-RM2 in patients scheduled for and/or undergoing wide local excision (WLE) with or without sentinel lymph node biopsy (SLNB) or complete axillary lymph node dissection(cALND) for breast cancer with an ER-positive invasive primary cancer.

The study consists of 3 sequential groups:

Group 1 (N=20 patients): Torso, i.e. base of skull to thighs, PET/CT imaging and axillary gamma probe measurements (using a collimator) of 68Ga-RM2 to: determine the optimal scan time-window post-injection; to extrapolate the optimal dose for resolution against axillary background signal on gamma probe measurements (first 6 patients); and the value of 68Ga-RM2 PET/CT imaging for breast cancer staging (all 20 patients).

Group 2 (N=10 patients): Intraoperative LightPath® imaging with 68Ga-RM2 to familiarise site with procedure and interpretation of intraoperative scans,validate the dose and timings determined from Group 1, and optimise LightPath® Imaging parameters such as acquisition resolution and duration. Group 2 scans will acquire LightPath® images of both intact and incised cancer specimens for post-operative standardised, controlled assessment. Group 2 will use the optimal scan time-window and 68Ga-RM2 activity extrapolated from at least the first 6 patients in Group 1. The dose of 68Ga-RM2 will be determined to optimise the intra-operative imaging and axillary gamma probe measurements.

Group 3 (N=50 patients): Intraoperative LightPath® imaging with 68Ga-RM2 to measure agreement between LightPath® images and post-operative histopathology. Group 3 scans will acquire LightPath® images of intact and incised cancer specimens for post-operative standardised, controlled assessment. Group 3 will use the optimal scan time-window and 68Ga-RM2 activity extrapolated from the first 6 patients in Group 1 with the optimised imaging parameters, and dose developed from Group 2.

The intraoperative LightPath® Images will be used to inform the surgeons about detectable residual cancer in an attempt to achieve better guided cancer surgery and complete tumour excision with clear WLE resection margins

The study site will use the local criteria considered standard of care to guide decisions to act on positive margins. Lightpoint Medical will provide guidance to act on LightPath® Images in the Instructions forUse (IFU). It will be at the Investigator's discretion to choose whether to act based upon the intraoperative LightPath® Images.

In Group 3,the resection margin status of the WLE specimen, cavity shavings (if any) and the metastatic status of axillary (sentinel) lymph nodes as measured with the LightPath® Imaging System will be compared with histopathology results. A positive margin on histology will be defined as

* Invasive carcinoma: positive: ink on tumour; close: <1mm; negative ≥1mm
* Ductal carcinoma in situ (DCIS)or pleomorphic lobular carcinoma in situ (LCIS) (if present): positive: ink on tumour; close: <2mm; negative ≥2mm.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have signed an informed consent form prior to any study related activity
* Subjects who are able to give voluntary, written informed consent to participate in this study.
* Subjects who are able to understand this study and are willing to complete all the study assessments
* Female subjects ≥18 years of age with a diagnosis of ER-positive invasive breast cancer. ER-positivity is defined as an Allred score of 3 or more on immunohistochemical analysis.
* Female subjects of childbearing age must have a negative pregnancy test (by Beta HCG qualitative analysis), or must have had a history of a surgical sterilisation, or must give history of no menses in the past twelve months
* Groups 2 and 3: Subjects scheduled for WLE +/-SLNB or ALND

Exclusion Criteria:

* Subjects who have had surgery in the operated breast in the past 12months
* Subjects who have had radiotherapy in the operated breast
* Subjects who have had neoadjuvant systemic therapy
* Subjects who have had systemic chemotherapy or investigational therapy in the past two years
* Subjects who are pregnant or lactating
* Subjects who have a known hypersensitivity to 68Ga, bombesin analogues, or GRPR-antagonists
* Subjects who have an existing medical condition that would compromise their participation in the study•Subjects with a current or active history of other known cancerin the opinion of the Investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-30 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of LightPath® Imaging System | up to 5 year
  Agreement between margin status determined by LightPath® Imaging and post-operative histopathology (Group 3)

SECONDARY OUTCOMES:
Optimal scan time-window for 68Ga-RM2 PET/CT imaging | 1 year
  Group 1 only
Gamma probe measurements (collimated) in the axilla to determine optimal 68Ga-RM2 activity | 1 year
  Group 1 only
Value of 68Ga-RM2 PET/CT imaging for breast cancer staging | 1 year
  Group 1 only
Radiation dosimetry measurements for the staff | 1 year
  Group 1 only
Optimal device settings, tracer dose, and working procedures | up to 2 years
  Group 2 only
Inter-rater agreement in post-operative standardised, controlled assessments of LightPath® Images | up to 5 year
  Group 3 only
MDT decision to re-operate at index location | up to 5 year
  Group 3 only
Weight of primary lump and lump plus shavings | up to 5 year
  Groups 2 and 3 only
Radiation dosimetry for operating room and recovery area staff | up to 5 year
  Groups 2 and 3 only

OTHER OUTCOMES:
Association between PET and/or LightPath® results and biomarkers (ER, PR, HER2, other according to local practice) | up to 5 year
  Exploratory Outcome Measures
Study-related adverse events (AEs) | up to 5 year
  Exploratory Outcome Measures
Lymph node involvement by LightPath® Image (compared with histology: macrometastasis, micrometastasis, or isolated tumour cells) | up to 5 year
  Exploratory Outcome Measures
Agreement between 68Ga-RM2 and gastrin-releasing peptide receptor (GRPR) immunohistochemistry | up to 5 year
  Exploratory Outcome Measures

CONTACTS AND LOCATIONS:
Overall Officials: Qamar B Akbar, MSc, Study Director — Lightpoint Medical Ltd
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No